CLINICAL TRIAL: NCT02025530
Title: The Midlands and North of England Stillbirth Study - A Case-Control Study of Modifiable Factors in Late Stillbirth
Brief Title: The Midlands and North of England Stillbirth Study
Acronym: MiNESS
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Alexander Heazell, Senior Clinical Lecturer in Obstetrics, University of Manchester
Other Study IDs: GN2156
Record Dates: First submitted 2013-12-20; First posted 2014-01-01 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Stillbirth
Keywords: Stillbirth; Modifiable risk factors
MeSH Terms: conditions — Stillbirth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Hair
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: A structured questionnaire will be administered to women who have experienced a late ≥ 28 weeks gestation stillbirth, who have a singleton pregnancy with no congenital abnormality.
  Interventions: Other: Questionnaire
- Controls: A structured questionnaire will be administered to controls. These are women matched to the case group by gestation and unit of birth, who have a normal ongoing singleton pregnancy with no congenital abnormality.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — An indepth interview will be carried out and a structured questionnaire will be completed by both cases and controls

SUMMARY:
The United Kingdom has one of the highest rates of stillbirth in Europe, with more than 4,000 stillbirths every year; which equates to more than 11 deaths every day. Furthermore, this rate has changed very little over the last 20 years. This loss of life and the adverse psychological consequences urgently needs addressing.

A recent New Zealand study investigating modifiable factors associated with stillbirth (the Auckland Stillbirth Study) found that mothers who did not go to sleep on their left side had a twofold risk of late stillbirth (≥28 weeks gestation) compared to mothers who did go to sleep on their left side. These novel findings need urgent confirmation.

This proposed study aims to confirm or refute these findings and to ascertain whether a preventative programme should be introduced. This proposed study aims to confirm or refute the findings of the Auckland Stillbirth Study.

Participants will be recruited from maternity units in the Midlands and North of England (led by centres in Liverpool, Manchester, West Yorkshire and Birmingham). 291 women with a singleton late stillbirth without congenital abnormality will be interviewed by research midwives shortly after the birth. A control group of 580 women with ongoing pregnancies will be interviewed at a gestation group matched to that at which stillbirths occurred. These data will determine whether an intervention study should be considered. If there is a causal relationship between maternal sleep position and late stillbirth we estimate that upto 37% of late stillbirths might be prevented.

DETAILED DESCRIPTION:
The death of an unborn child is a prevalent and tragic public health problem which currently affects millions of families worldwide. Late stillbirth (at or beyond 28 weeks of gestation) is one of the few potentially avoidable maternal and child health problems where the rate of decline in high income countries has slowed in recent decades [1]. The United Kingdom currently has one of the highest rates of stillbirth in Europe, ranking 33rd out of 35 high income countries.

The variations in stillbirth rates between high income countries suggest that it should be possible to make further reductions in late stillbirths. The estimated annual reduction in rates of late stillbirth over recent decades is about 1.1% [1], compared to 2.1% for neonatal death rates, with a resultant increase in the proportion of perinatal deaths (stillbirths plus neonatal deaths) attributable to stillbirth [2]. The Lancet Stillbirth Series [1, 3, 4] has highlighted the silent but prevalent public health problem of stillbirth and together with Sands and the Royal College Of Obstetricians and Gynaecologists has called for research to address these unacceptably high rates.

Current established risk factors for late stillbirth in high income countries include: advanced maternal age (>35 years) [5], high pre-pregnancy body mass index (BMI) [6], smoking [7], reduced antenatal care attendance [8], low socioeconomic status [8] and small for gestational age (SGA) infants [9]. A meta-analysis of population based studies addressing risk factors for stillbirth found that the three most important modifiable risk factors were overweight and obesity (population attributable risk 818%) advanced maternal age (population attributable risk 68%), and smoking (population attributable risk 47%) [3]. Of these only, cigarette smoking may be realistically addressed after pregnancy has started. There has been limited research investigating the role of novel, modifiable factors which have the potential to advance knowledge and address the important gaps in the field of stillbirth research.

This study aims to explore modifiable risk factors for late stillbirth in the UK and to substantiate the recent identification of a new modifiable risk factor for unexpected late pregnancy stillbirths. In the Auckland Stillbirth Study [10] our New Zealand collaborators discovered an approximately two-fold increase in late stillbirth with non-left sided maternal sleep position on the night before the baby died. In addition, women who did not get up at night and those who slept during the day were also at increased risk of stillbirth. The strength of this primary finding was unanticipated and now maternal sleep position requires urgent, rigorous evaluation in another population. MiNESS aims to address these factors.

This multi-centered case control study will recruit 291 women who have experienced a late (≥28 weeks gestation) matched with 580 women who have a continuing pregnancy at the same gestation (controls). The women will be interviewed by an experienced research midwife and an in depth questionnaire will be completed.

Analysis will be carried out using the standard Mantel-Haenszel odds ratio analysis used in case-control studies. Unconditional logistic regression will be used to adjust for potential confounders and to determine the presence of interactions.

ELIGIBILITY:
Inclusion Criteria: CASES

* Women who experience a stillbirth ≥28 weeks gestation in a participating unit.

Exclusion Criteria:

* Fetal death prior to 28 weeks gestation.
* Women who's babies have a significant congenital abnormality.
* Women with multiple pregnancy.
* Maternal age below 16 years.
* Women unable to give informed consent.

Inclusion Criteria: CONTROLS

* Women with a normal pregnancy matched to gestation and unit of birth to the cases.

Exclusion Criteria:

* Pregnancy under 28 weeks gestation.
* Women who's babies have a significant congenital abnormality.
* Women with multiple pregnancy.
* Maternal age below 16 years.
* Women unable to give informed consent.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample will be recruited from maternity units in the Midlands and the North of England.
Sampling Method: Probability Sample
Enrollment: 1030 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasina Stacey, Principal Investigator — Mid Yorkshire NHS Trust; Edwin Mitchell, Principal Investigator — University of Auckland, New Zealand; Lesley McCowan, Principal Investigator — University of Auckland, New Zealand; Bill Martin, Principal Investigator — Birmingham Women's Hospital NHS Foundation Trust; Devender Roberts, Principal Investigator — Liverpool Women's NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Liverpool Women's NHS Foundation Trust, Liverpool, Merseyside
  - Birmingham Women's Hospital NHS Foundation Trust, Birmingham, West Midlands
  - Mid Yorkshire NHS Trust, Dewsbury, Yorkshire
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester

REFERENCES:
- [Background] Cousens S, Blencowe H, Stanton C, Chou D, Ahmed S, Steinhardt L, Creanga AA, Tuncalp O, Balsara ZP, Gupta S, Say L, Lawn JE. National, regional, and worldwide estimates of stillbirth rates in 2009 with trends since 1995: a systematic analysis. Lancet. 2011 Apr 16;377(9774):1319-30. doi: 10.1016/S0140-6736(10)62310-0. PMID 21496917
- [Background] Rajaratnam JK, Marcus JR, Flaxman AD, Wang H, Levin-Rector A, Dwyer L, Costa M, Lopez AD, Murray CJ. Neonatal, postneonatal, childhood, and under-5 mortality for 187 countries, 1970-2010: a systematic analysis of progress towards Millennium Development Goal 4. Lancet. 2010 Jun 5;375(9730):1988-2008. doi: 10.1016/S0140-6736(10)60703-9. Epub 2010 May 27. PMID 20546887
- [Background] Flenady V, Koopmans L, Middleton P, Froen JF, Smith GC, Gibbons K, Coory M, Gordon A, Ellwood D, McIntyre HD, Fretts R, Ezzati M. Major risk factors for stillbirth in high-income countries: a systematic review and meta-analysis. Lancet. 2011 Apr 16;377(9774):1331-40. doi: 10.1016/S0140-6736(10)62233-7. PMID 21496916
- [Background] Froen JF, Cacciatore J, McClure EM, Kuti O, Jokhio AH, Islam M, Shiffman J; Lancet's Stillbirths Series steering committee. Stillbirths: why they matter. Lancet. 2011 Apr 16;377(9774):1353-66. doi: 10.1016/S0140-6736(10)62232-5. PMID 21496915
- [Background] Rasmussen S, Albrechtsen S, Irgens LM, Dalaker K, Maartmann-Moe H, Vlatkovic L, Markestad T. Risk factors for unexplained antepartum fetal death in Norway 1967-1998. Early Hum Dev. 2003 Feb;71(1):39-52. doi: 10.1016/s0378-3782(02)00111-1. PMID 12614949
- [Background] Stephansson O, Dickman PW, Johansson A, Cnattingius S. Maternal weight, pregnancy weight gain, and the risk of antepartum stillbirth. Am J Obstet Gynecol. 2001 Feb;184(3):463-9. doi: 10.1067/mob.2001.109591. PMID 11228504
- [Background] Wisborg K, Kesmodel U, Henriksen TB, Olsen SF, Secher NJ. Exposure to tobacco smoke in utero and the risk of stillbirth and death in the first year of life. Am J Epidemiol. 2001 Aug 15;154(4):322-7. doi: 10.1093/aje/154.4.322. PMID 11495855
- [Background] Huang DY, Usher RH, Kramer MS, Yang H, Morin L, Fretts RC. Determinants of unexplained antepartum fetal deaths. Obstet Gynecol. 2000 Feb;95(2):215-21. doi: 10.1016/s0029-7844(99)00536-0. PMID 10674582
- [Background] Cnattingius S, Haglund B, Kramer MS. Differences in late fetal death rates in association with determinants of small for gestational age fetuses: population based cohort study. BMJ. 1998 May 16;316(7143):1483-7. doi: 10.1136/bmj.316.7143.1483. PMID 9582131
- [Background] Stacey T, Thompson JM, Mitchell EA, Ekeroma AJ, Zuccollo JM, McCowan LM. Association between maternal sleep practices and risk of late stillbirth: a case-control study. BMJ. 2011 Jun 14;342:d3403. doi: 10.1136/bmj.d3403. PMID 21673002
- [Derived] Budd J, Stacey T, Martin B, Roberts D, Heazell AEP. Women's experiences of being invited to participate in a case-control study of stillbirth - findings from the Midlands and North of England Stillbirth Study. BMC Pregnancy Childbirth. 2018 Aug 6;18(1):317. doi: 10.1186/s12884-018-1956-1. PMID 30081858
- [Derived] Heazell AEP, Budd J, Li M, Cronin R, Bradford B, McCowan LME, Mitchell EA, Stacey T, Martin B, Roberts D, Thompson JMD. Alterations in maternally perceived fetal movement and their association with late stillbirth: findings from the Midland and North of England stillbirth case-control study. BMJ Open. 2018 Jul 6;8(7):e020031. doi: 10.1136/bmjopen-2017-020031. PMID 29982198
- [Derived] Platts J, Mitchell EA, Stacey T, Martin BL, Roberts D, McCowan L, Heazell AE. The Midland and North of England Stillbirth Study (MiNESS). BMC Pregnancy Childbirth. 2014 May 21;14:171. doi: 10.1186/1471-2393-14-171. PMID 24885461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between April 2014 and March 2016 from 41 maternity units around the United Kingdom.
Pre-assignment Details: This was a case-control study, so participants were not assigned to a specific arm/group. 5 cases (women who had a stillbirth) were excluded prior to analysis because the baby was found to have a congenital anomaly at post-mortem examination. One control (women with a live baby at interview) was excluded because she had a stillborn baby.
Groups:
- Cases: A structured questionnaire was administered to women who have experienced a late ≥ 28 weeks gestation stillbirth, who have a singleton pregnancy with no congenital abnormality.
  Questionnaire: An indepth interview will be carried out and a structured questionnaire will be completed by both cases and controls.
  Clinical information was obtained from maternal case notes following the interview.
- Controls: A structured questionnaire was administered to controls. These are women matched to the case group by gestation and unit of birth, who have a normal ongoing singleton pregnancy with no congenital abnormality.
  Questionnaire: An indepth interview will be carried out and a structured questionnaire will be completed by both cases and controls.
  Clinical information was obtained from maternal case notes following the interview.
Period: Overall Study
Arm/Group | Cases | Controls
Started | 296 | 734
Completed | 291 | 733
Not Completed | 5 | 1
Not completed — No longer met elligibility criteria | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cases (Stillbirth): A structured questionnaire was administered to women who have experienced a late ≥ 28 weeks gestation stillbirth, who have a singleton pregnancy with no congenital abnormality.
  Questionnaire: An indepth interview will be carried out and a structured questionnaire will be completed by both cases and controls.
  Clinical information was obtained from maternal case notes following the interview.
- Controls (Live Pregnancy): A structured questionnaire was administered to controls. These are women matched to the case group by gestation and unit of birth, who have a normal ongoing singleton pregnancy with no congenital abnormality.
  Questionnaire: An indepth interview will be carried out and a structured questionnaire will be completed by both cases and controls.
  Clinical information was obtained from maternal case notes following the interview.
- Total: Total of all reporting groups
Arm/Group | Cases (Stillbirth) | Controls (Live Pregnancy) | Total
Number analyzed (Participants) | 291 | 733 | 1024
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (5.9) | 30.4 (5.1) | 30.3 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291 | 733 | 1024
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maternal Sleep Practices During Pregnancy
Description: Self-reported going to sleep position in late pregnancy
Time Frame: One night prior to questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Cases (Stillbirth) | Controls (Live Pregnancy)
Number analyzed (Participants) | 291 | 733
Participants
  Left | 140 | 383
  Right | 73 | 220
  Back | 19 | 24
  Tummy | 3 | 4
  Propped | 9 | 15
  Variable | 32 | 76
  Unknown | 15 | 11

2. Secondary Outcome: Maternal Perception of Fetal Activity
Description: Maternal Perception of Fetal Activity reported via the researcher-administered questionnaire.
Time Frame: Two weeks prior to stillbirth / interview
Measure: Count of Participants; unit: Participants
Arm/Group | Cases (Stillbirth) | Controls (Live Pregnancy)
Number analyzed (Participants) | 291 | 733
Participants
  In last 2 weeks did movements increase? | 37 | 254
  In last 2 weeks did movements decrease? | 86 | 63
  Movements stayed the same | 153 | 397
  Unsure | 15 | 19

3. Post Hoc Outcome: Screening for Gestational Diabetes and Fasting Plasma Glucose
Description: Performance of 75g oral glucose tolerance test and the results of glucose tolerance test in cases and controls
Time Frame: During index pregnancy
Population: Women were excluded from this analysis if they had pre-existing diabetes. Women should have been screened using oral glucose tolerance test if they had a positive family history, were of South Asian or Black Caribbean ethnicity, had a body mass index ≥ 30 kg/m2, or previous pregnancy effected by GDM or macrosomic (birthweight ≥4.5 kg) birth.
Measure: Count of Participants; unit: Participants
Arm/Group | Cases (Stillbirth) | Controls (Live Pregnancy)
Number analyzed (Participants) | 283 | 729
Participants
  Women screened by Oral Glucose Tolerance Test | 94 | 277
  Proportion Diagnosed with GDM | 6 | 30

ADVERSE EVENTS:
Time Frame: For the duration of participation in the study (e.g. from recruitment until pregnancy outcome for participants in the control arm). As this was an observational study no SAEs were attributed to completion of the maternal questionnaire.
Description: Stillbirth was not recorded as an adverse event in the case group because it was an entry criteria for the study.
Arm/Group | Cases (Stillbirth) | Controls (Live Pregnancy)
All-Cause Mortality (participants affected / at risk) | 0/296 | 0/734
Serious Adverse Events (participants affected / at risk) | 0/296 | 0/734
Other Adverse Events (participants affected / at risk) | 0/296 | 0/734

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes